CLINICAL TRIAL: NCT01711060
Title: A Comparison of Balloon Catheter Versus Ocytocin for Cervical Ripening on Scarred Uterus With Unfavorable Cervix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CICATAC
Record Dates: First submitted 2012-08-23; First posted 2012-10-22 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Scarred Uterus
MeSH Terms: interventions — Oxytocin

ARMS (2):
- oxytocin (Experimental)
  Interventions: Drug: oxytocin
- balloon catheter (Experimental): Dufour 1859H18
  Interventions: Procedure: balloon catheter

INTERVENTIONS:
Drug: oxytocin
  Arms: oxytocin
Procedure: balloon catheter
  Arms: balloon catheter

SUMMARY:
Increasing cesarean rate in France is worrying. Different methods are described for ripening labor : the use of prostaglandins is described but maybe dangerous for patients with scarred uterus and is not recommended.

Intracervical balloon is an efficient alternative methods which as already been tested for unfavorable cervix ripening on nulliparous women.

But it was rarely tested on women with scared uterus and unfavorable cervix (bishop score <4).

The investigators propose a prospective randomised trial comparing cervix ripening with intracervical balloon inflated by 50 ml sterile water during 12 hours versus ocytocin (reference method).

The investigators expect to demonstrate what it's a safe method to increase vaginal delivery for women with previous cesarean section who need an induction of labour.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy over 37 weeks
* Singleton pregnancy
* Vertex presentation
* Previous caesarean section with unique Transversal segmentary incision
* Medical indication of induction of labor
* Unfavorable cervix with Bishop score < 4
* No Premature Rupture Of Membranes
* Informed consent

Exclusion Criteria:

* Before 18 years old
* Placenta Praevia
* Premature Rupture Of Membranes
* Uterine scar other than transversal segmentary incision
* Cervical infection (except Streptoccoccus Agalactiae carrier) or choriamnionitis
* Multiple pregnancy
* Fetal malpresentation
* Cesarean indication
* Latex allergy
* No informed consent

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2010-12; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Rate of childbirth by low way
  The childbirth by low way being considered as a success of the treatment

SECONDARY OUTCOMES:
Rate of incidence of materno-fœtales morbidity
  number

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Service Gynécologie Obstétrique, Angoulême
  - Service Gynécologie Obstétrique, Bressuire
  - Service Gynécologie Obstétrique, Châtellerault
  - Service Gynécologie Obstétrique, Nancy
  - Service Gynécologie Obstétrique et médecine de la reproduction, Poitiers
  - Service Gynécologie Obstétrique, Rennes
  - Service Gynécologie Obstétrique, Toulouse

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264